CLINICAL TRIAL: NCT04526964
Title: Improved Health Care for People With Chronic Heart Disease and Implanted Cardiac Support Through Curricular Self-management - Phase 3: Randomized Controlled Trial (RCT)
Brief Title: Improved Self-management for Patients on Ventricular Assist Device (VAD) Support - Phase 3
Acronym: SELMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Freiburg (Other)
Collaborators: University Heart Center Freiburg - Bad Krozingen (Other); Heart and Diabetes Center North Rhine-Westphalia (Other); German Heart Center (Other); Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Christiane Kugler, Professor Doctor. rer. biol. hum., University of Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01VSF18012 (Phase 3)
Record Dates: First submitted 2020-08-14; First posted 2020-08-26 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Ventricular Assist Device; Psychosocial Factors; Self-management
Keywords: Ventricular Assist Device; Psychosocial Factors; Evidence-based Curriculum; Self-management

STUDY DESIGN:
Intervention Model Description: This RCT will be conducted at four established cardiac centers in Germany. Participants will be assigned to either intervention or control using a 1: 1 randomization scheme. Block-randomization will be performed by a professional from the study coordinating center not being involved into the clinical care for patients. The group assignment is non-blinded to the professionals involved in order to enable the intervention to be carried out adequately. Participants in the control group (CGr) receive standard follow-up procedures (care as usual). The intervention group (IGr) receive self-management support and skills training based on the modular self-management curriculum post-implant and during regular outpatient follow-up. The self-management training program will be supplemented by a smartphone-based application. The intervention lasts for 3 months followed by a 9-month follow-up period per participant. Based on power calculations the inclusion of 142 patients is anticipated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IGr) (Other): Participants of the intervention group (IGr) receive self-management support and skills training based on the modular self-management curriculum during the inpatient post-implant phase, as well as one refresher session about six weeks after discharge during regular outpatient follow-up and a supplementary app.
  Interventions: Behavioral: Self-management curriculum
- Control Group (CGr) (No Intervention): Participants in the control group (CGr) receive the standard follow-up procedures (care as usual).

INTERVENTIONS:
Behavioral: Self-management curriculum — The Intervention starts during inpatient phase after relocation of potential study participants from the intensive care unit to normal ward and after informed consent to participate. Those subjects assigned to the CGr by randomization code receive standard care at the respective center. Subjects assigned to the IGr received, in addition to standard care, a multi-modular self-management training carried out at the respective center. The content of the self-management training should be deepened and consolidated through a supplementary app. Training is performed during inpatient post-implant phase, as well as one refresher session about six weeks after discharge during regular outpatient follow-up. The intervention lasts 3 months, plus a 9-month follow-up per subject. The content of the self-management training is based on current evidence and was written in a curriculum to achieve the highest possible standardization, taking into account the center specifics.
  Arms: Intervention Group (IGr)

SUMMARY:
The number of patients suffering from end-stage heart disease challenges healthcare services in the western world, where an estimated 1-2% of the population suffer from this chronic condition. Ventricular assist device (VAD) implantations have become a common therapeutic strategy for those affected. Live with a VAD, however, is far from normal and does expose patients to multiple challenges and the need to adjust to a complex self-management. Inadequate self-management can lead to serious complications, specifically neuro-cognitive events, bleeding, and exit-site related wound infections may impair the outcome following the VAD implantation procedure.

Based on systematized literature review and a previous prevalence assessment study (ClinicalTrials.gov Identifier: NCT04234230), a modular evidence-based curriculum has been developed by a multiprofessional group of experts. This curriculum aims at improving knowledge, skills, and competencies for those affected to empower VAD patients to better self-manage their everyday life with the VAD, and to regain quality of life. This study focuses on a multi-center implementation and evaluation of the curriculum using a fully powered randomized-controlled study (RCT) design. This RCT will be conducted at four established cardiac centers throughout Germany. Participants will be assigned to either intervention or control using a 1: 1 randomization scheme. Block-randomization will be performed by a professional from the study coordinating center not being involved into the clinical care for patients. At the participating sites, the group assignment is non-blinded to the professionals involved in order to enable the intervention so be carried out adequately. Participants in the control group (CGr) receive the standard follow-up procedures (care as usual). Participants in the intervention group (IGr) receive self-management support and skills training based on the modular self-management curriculum post-implant, and during regular outpatient follow-up. The intervention lasts for 3 months followed by a 9-month follow-up per participant. Based on the power calculations the inclusion of 142 patients is anticipated.

DETAILED DESCRIPTION:
The number of patients suffering from end-stage heart disease challenges healthcare services in the western world, where an estimated 1-2% of the population suffer from this chronic condition. Ventricular assist device (VAD) implantations have become a common therapeutic strategy for those affected. Indications include a multi-year bridging therapy (up to 10 years) and increasingly a destination therapy. The Euromacs Registry published the second report in 2018 and reported 2,947 registered VAD implantations in 2016 (+257 percent). Euromacs further points to a rising trend and demand for the use of VAD systems for the treatment of patients with end-stage failure (NYHA classes III and IV). In Germany, an increase of VAD implantation by 36.6 percent has been reported since 2011. The position paper of the German Society of Cardiology (2016) warns that the range of indications for VAD implantation for people with chronic heart disease will continue to change. The ISHLT Guideline (International Society for Heart and Lung Transplantation), published in 2018, calls for psychosocial care and standardized self-management skills of patients before, during and in the long-term after VAD implantation. This is currently being implemented inconsistently in terms of structure and quality in German cardiac centers. Live with a VAD, however, is far from normal and does expose patients to multiple challenges and the need to adjust to a complex self-management. Inadequate self-management can lead to serious complications, specifically neuro-cognitive events, bleeding, and exit-site related wound infections may impair the outcome following the VAD implantation procedure.

The design for this study will be a fully-powered block-randomized trial (RCT). This RCT will be conducted at four established cardiac centers throughout Germany. Participants will be assigned to either intervention or control using a 1: 1 randomization scheme. Block-randomization will be performed by a professional from the study coordinating center not being involved into the clinical care for patients. At the participating sites, the group assignment is non-blinded to the professionals involved in order to enable the intervention so be carried out adequately. Participants in the control group (CGr) receive the standard follow-up procedures (care as usual). Participants in the intervention group (IGr) receive self-management support and skills training based on the modular self-management curriculum post-implant, and during regular outpatient follow-up. The self-management training program will be supplemented by a smartphone-based application. The smartphone application will be downloaded optionally on the patients' own smartphones, and patients will be instructed on how to use it. In the app, the study participants can receive additional information on health-related data, e.g. weight, temperature, sleep or mood. Entering health related data is absolutely voluntary. No data will be transferred to the clinical sites. The study participants can also use the app to read VAD related information only without any registration. Data entered (optional) are used only for the participants' own information overview. The intervention lasts for 3 months followed by a 9-month follow-up period per participant. Based on the power calculations the inclusion of 142 patients is anticipated.

The expected results can improve self-management, self-efficacy, and health-related quality of life for patients on VAD support. In addition, a reduction in VAD-specific complications and inpatient admission rates due to reduced complication rates can expected. The project aims to improve long-term psychosocial care through self-management support for patients on VAD support. The modular curriculum and the supporting

ELIGIBILITY:
Inclusion Criteria:

* Stable postoperative condition
* Outpatient treatment at the respective heart center
* 18 years and older
* No contraindications (e.g. Cognitive, Language)
* Signed Informed Consent

Exclusion Criteria:

* Not an outpatient at the respective heart center
* Underage
* Contraindications (e.g. Cognitive, Language)
* No signed Informed Consent
* Participation in other behavior-related studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Self-management Skills from 2-4 Weeks Post-implant (T1) to 12 Months Post-implant (T3) | From 2-4 weeks post-implant to 12 months post-implant
  Self-managment skills and needs of the participants (for example medication intake or infection prevention) measured with a self-assessment questionnaire ("SELMA questionnaire").

SECONDARY OUTCOMES:
Change in Health-related Quality of Life From 2-4 Days Post-implant (T0) to 12 Months Post-implant (T3) | From 2-4 days post-implant to 12 months post-implant
  The perceived health-related quality of life of the participants measured with the self-assessment questionnaire "QoL-VAD". Values range from 0 to 100 for each scale with higher values indicate better outcome.
Change in Perceived Social Support From 2-4 Weeks Post-implant (T1) to 12 Months Post-implant (T3) | From 2-4 weeks post-implant to 12 months post-implant
  The perceived social support of the participants measured with the brief form of the "Perceived Social Support Questionnaire" (F-SozU K-14). Higher scores indicate better outcomes.
Change in Symptoms of Anxiety From 2-4 Days Post-implant (T0) to 12 Months Post-implant (T3) | From 2-4 days post-implant to 12 months post-implant
  Symptoms of anxiety measured with the screening instrument "Hospital Anxiety and Depression Scale" (HADS). Values range from 0 to 21 for each scale with higher values indicate worse outcome.
Change in Symptoms of Depression From 2-4 Days Post-implant (T0) to 12 Months Post-implant (T3) | From 2-4 days post-implant to 12 months post-implant
  Symptoms of depression measured with the screening instrument "Hospital Anxiety and Depression Scale" (HADS). Values range from 0 to 21 for each scale with higher values indicate worse outcome.
Change in Adverse Event Rates From 2-4 Days Post-implant (T0) to 12 Months Post-implant (T3) | From 2-4 days post-implant to 12 months post-implant
  Potentially relevant adverse events, the number of neurocognitive events, the number of bleeding events, and the number of and exit-site related wound infections will be taken from the medical record of the participants.

OTHER OUTCOMES:
Change in Comorbidities From 2-4 Days Post-implant (T0) to 12 Months Post-implant (T3) | From 2-4 days post-implant to 12 months post-implant
  Relevant comorbidities (e.g. Diabetes, Hypertension, psychic comorbidities) will be taken from the medical record of the participants.
VAD Type | 2-4 days post-implant
  Information on implanted VAD type (HVAD, HMIII or other) will be taken from the medical record of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Kugler, Prof. Dr., Study Director — University of Freiburg
Locations (4):
- Germany (4):
  - University Heart Center Freiburg • Bad Krozingen, Freiburg im Breisgau, Baden-Wurttemberg
  - Heart and Diabetes Center NRW, Bad Oeynhausen, Bad Oeynhausen, North Rhine-Westphalia
  - Leipzig Heart Center, Leipzig, Saxony
  - German Heart Center Berlin, Berlin

REFERENCES:
- [Background] Feldman D, Pamboukian SV, Teuteberg JJ, Birks E, Lietz K, Moore SA, Morgan JA, Arabia F, Bauman ME, Buchholz HW, Deng M, Dickstein ML, El-Banayosy A, Elliot T, Goldstein DJ, Grady KL, Jones K, Hryniewicz K, John R, Kaan A, Kusne S, Loebe M, Massicotte MP, Moazami N, Mohacsi P, Mooney M, Nelson T, Pagani F, Perry W, Potapov EV, Eduardo Rame J, Russell SD, Sorensen EN, Sun B, Strueber M, Mangi AA, Petty MG, Rogers J; International Society for Heart and Lung Transplantation. The 2013 International Society for Heart and Lung Transplantation Guidelines for mechanical circulatory support: executive summary. J Heart Lung Transplant. 2013 Feb;32(2):157-87. doi: 10.1016/j.healun.2012.09.013. No abstract available. PMID 23352391
- [Background] de By TMMH, Mohacsi P, Gahl B, Zittermann A, Krabatsch T, Gustafsson F, Leprince P, Meyns B, Netuka I, Caliskan K, Castedo E, Musumeci F, Vincentelli A, Hetzer R, Gummert J; EUROMACS members. The European Registry for Patients with Mechanical Circulatory Support (EUROMACS) of the European Association for Cardio-Thoracic Surgery (EACTS): second report. Eur J Cardiothorac Surg. 2018 Feb 1;53(2):309-316. doi: 10.1093/ejcts/ezx320. PMID 29029117
- [Background] de By TM, Mohacsi P, Gummert J, Bushnaq H, Krabatsch T, Gustafsson F, Leprince P, Martinelli L, Meyns B, Morshuis M, Netuka I, Potapov E, Zittermann A, Delmo Walter EM, Hetzer R; EUROMACS members. The European Registry for Patients with Mechanical Circulatory Support (EUROMACS): first annual report. Eur J Cardiothorac Surg. 2015 May;47(5):770-6; discussion 776-7. doi: 10.1093/ejcts/ezv096. Epub 2015 Mar 27. PMID 25820161
- [Background] Beckmann A, Funkat AK, Lewandowski J, Frie M, Ernst M, Hekmat K, Schiller W, Gummert JF, Cremer JT. Cardiac Surgery in Germany during 2014: A Report on Behalf of the German Society for Thoracic and Cardiovascular Surgery. Thorac Cardiovasc Surg. 2015 Jun;63(4):258-69. doi: 10.1055/s-0035-1551676. Epub 2015 May 26. PMID 26011675
- [Background] Reichenspurner H. Geleitwort zu "Rehabilitationsstandards fur die Anschlussheilbehandlung und allgemeine Rehabilitation fur Patienten mit einem Herzunterstutzungssystem (VAD Ventricular Assist Device)". Clin Res Cardiol Suppl. 2016 Mar;11 Suppl 1:1. doi: 10.1007/s11789-016-0080-x. No abstract available. German. PMID 26882904
- [Background] Dew MA, DiMartini AF, Dobbels F, Grady KL, Jowsey-Gregoire SG, Kaan A, Kendall K, Young QR, Abbey SE, Butt Z, Crone CC, De Geest S, Doligalski CT, Kugler C, McDonald L, Ohler L, Painter L, Petty MG, Robson D, Schloglhofer T, Schneekloth TD, Singer JP, Smith PJ, Spaderna H, Teuteberg JJ, Yusen RD, Zimbrean PC. The 2018 ISHLT/APM/AST/ICCAC/STSW recommendations for the psychosocial evaluation of adult cardiothoracic transplant candidates and candidates for long-term mechanical circulatory support. J Heart Lung Transplant. 2018 Jul;37(7):803-823. doi: 10.1016/j.healun.2018.03.005. Epub 2018 Apr 27. PMID 29709440
- [Background] Kato N, Jaarsma T, Ben Gal T. Learning self-care after left ventricular assist device implantation. Curr Heart Fail Rep. 2014 Sep;11(3):290-8. doi: 10.1007/s11897-014-0201-0. PMID 24831883
- [Background] Eshelman AK, Mason S, Nemeh H, Williams C. LVAD destination therapy: applying what we know about psychiatric evaluation and management from cardiac failure and transplant. Heart Fail Rev. 2009 Mar;14(1):21-8. doi: 10.1007/s10741-007-9075-5. Epub 2008 Jan 24. PMID 18214674
- [Background] Kugler C, Bara C, von Waldthausen T, Einhorn I, Haastert B, Fegbeutel C, Haverich A. Association of depression symptoms with quality of life and chronic artery vasculopathy: a cross-sectional study in heart transplant patients. J Psychosom Res. 2014 Aug;77(2):128-34. doi: 10.1016/j.jpsychores.2014.06.007. Epub 2014 Jun 23. PMID 25077854
- [Background] Kugler C, Meng M, Rehn E, Morshuis M, Gummert JF, Tigges-Limmer K. Sexual activity in patients with left ventricular assist devices and their partners: impact of the device on quality of life, anxiety and depression. Eur J Cardiothorac Surg. 2018 Apr 1;53(4):799-806. doi: 10.1093/ejcts/ezx426. PMID 29211843
- [Background] Caro MA, Rosenthal JL, Kendall K, Pozuelo L, Funk MC. What the Psychiatrist Needs to Know About Ventricular Assist Devices: A Comprehensive Review. Psychosomatics. 2016 May-Jun;57(3):229-37. doi: 10.1016/j.psym.2016.01.002. Epub 2016 Jan 12. PMID 27005723
- [Derived] Kugler C, Spielmann H, Seemann M, Lauenroth V, Wacker R, Albert W, Spitz-Koeberich C, Semmig-Koenze S, von Cube M, Tigges-Limmer K. Self-management for patients on ventricular assist device support: a national, multicentre study: protocol for a 3-phase study. BMJ Open. 2021 May 5;11(5):e044374. doi: 10.1136/bmjopen-2020-044374. PMID 33952544